CLINICAL TRIAL: NCT07115615
Title: Exploring the Efficacy of Accelerated Transcranial Direct Current Stimulation (tDCS) as Adjunct to Pharmacotherapy in the Treatment of Obsessive-compulsive Disorder: A Randomized Controlled Trial Using High-resolution MRI
Brief Title: Exploring the Efficacy of Accelerated Transcranial Direct Current Stimulation (tDCS) as Adjunct to Pharmacotherapy in the Treatment of Obsessive-compulsive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Qing ZHAO, Attending Physician, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-YG-OCD
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Obsessive Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Active Comparator): Cathode transcranial direct current stimulation over the right OFC will be applied four times a day (2 hours interval), 5 days a week, for 1 week.
  Interventions: Device: high-definition transcranial direct current stimulation
- sham tDCS (Sham Comparator): The sham transcranial direct current stimulation over the right OFC will be applied four times a day (2 hours interval), 5 days a week, for 1 week.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: high-definition transcranial direct current stimulation — The tDCS device will deliver a direct current of 2mA during 20 minutes. Cathode electrode will be localized in front of the right OFC on the Fp2 point according to the EEG international reference. Four anode electrodes will be placed around FP2 (i.e. Fpz, AFz, AF4, AF8)
  Arms: active tDCS
Device: Sham tDCS — To demonstrate the same stimulation sensation as under real conditions, only 40 seconds of real stimulation (2mA) are given at the beginning of the treatment. In the remaining 20 minutes, only about 15ms of short current pulses of 110uA occur every 550ms.
  Arms: sham tDCS

SUMMARY:
This study will evaluate the decision-making ability and therapeutic effects of accelerated Transcranial Direct Current Stimulation (tDCS) as adjunct to pharmacotherapy in obsessive-compulsive disorder (OCD) patients, and the underlying neural mechanism by EEG and MRI.

DETAILED DESCRIPTION:
The purpose of this study is to examine the decision-making ability and clinical efficacy of accelerated tDCS over orbitofrontal cortex (OFC) as adjunct to pharmacotherapy in treatment of OCD patients.60 OCD patients on stable medication will be randomized into two groups (i.e. active or sham stimulation). Accelerated tDCS stimulation will be performed four times a day, five times a week, for one week. Iowa Gambling Task will be conducted at the baseline, after the one week tDCS and at the 1-month follow-up to evaluate the decision-making ability of OCD patients.The investigators will assess symptom severity before and after one week of tDCS. Through the study, Yale-Brown Obsessive Compulsive Scale（Y-BOCS）, Clinical Global Impression(CGI), the Obsessive Compulsive Inventory-Revised (OCI-R), the Beck Depression Inventory-II (BDI-II), the Beck Anxiety Inventory (BAI), Childhood Trauma Questionnair(CTQ), side-effect questionnaire and other scales will be obtained by a trained investigator.The patients will also receive magnetic resonance imaging (MRI) scan, electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old, Han ethnicity, right-handed
2. DSM-5 criteria for OCD;
3. Y-BOCS total score ≥16, receiving stable medication for at least 4 weeks before tDCS stimulation.
4. Years of education ≥9.

Exclusion Criteria:

1. Any axis I psychiatric disorder comorbidity
2. Severe obsessive-compulsive symptoms that render the patient unable to complete required assessment procedures.
3. Previous treatment with electroconvulsive therapy (ECT), repetitive transcranial magnetic stimulation (rTMS), or transcranial direct current stimulation (tDCS).
4. Severe somatic diseases or any physical conditions that may induce epilepsy or intracranial hypertension, including cardiovascular and respiratory diseases, etc.
5. History of neurological disorders (e.g., epilepsy, cerebrovascular accidents) or traumatic brain injury/brain surgery.
6. Implantation of intracranial stents, cardiac pacemakers, coronary stents, cochlear implants, or other internal medical devices.
7. Women who are pregnant or planning to become pregnant in the near future.
8. Serious suicide risks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement assessed by the Yale-Brown Obsessive Compulsive Scale(Y-BOCS) | Up to 5 weeks
  The responder on Y-BOCS is defined as a Y-BOCS decrease at least 35% from the baseline at post-treatment.

SECONDARY OUTCOMES:
The Beck Depression Inventory-II(BDI-II) | Up to 5 weeks
  It is a 21-item self-report measure scored on a 4-point Likert-type scale to summarize recent symptoms of depression.
The Beck Anxiety Inventory (BAI) | Up to 5 weeks
  It is a 21-item self-report inventory that is used for measuring the severity of anxiety.
Side-effect questionnaire | Up to 5 weeks
  It consists of ten commonly-reported side effects as well as an "other" category that allows participants to describe experiences/sensations not otherwise covered to rate the intensity of side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China